CLINICAL TRIAL: NCT02010684
Title: University of California, Los Angeles (UCLA)/Drew Project EXPORT: Mood and Diabetes Empowerment & Improvement Training (MADE IT)
Brief Title: Mood and Diabetes Empowerment & Improvement Training
Acronym: MADE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Dr. Jeanne Miranda, Jeanne Miranda Ph.D., University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MADE-IT Study 1P20MD00148-03
Record Dates: First submitted 2013-08-01; First posted 2013-12-13 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Depression; Self care; Empowerment; Behavioral intervention; Cognitive behavioral therapy; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Depression; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait-listed Control Group (No Intervention): Participants in the Wait-listed Control Group will receive augmented access and communication with a primary care provider. The augmentation would consist of providing the participant with a letter to be shared with their primary care doctor indicating their Hb A1c level and depression score at the time of eligibility screening. The research team will also attach a list of local mental health service providers to the letter. The participants randomized to the wait-listed control group will also be offered access to the intervention after the trial is completed in the event that the randomized controlled trial (RCT) has significant results.
- Empowerment and CBT Classes (Experimental): Participants will attend weekly 2-hour group Empowerment and CBT classes for 12 weeks led by two trained health educators. Participants will learn cognitive behavioral therapy (CBT) techniques to manage their mood. After CBT, participants will learn a diabetes education format that is grounded in empowerment theory that employs group problem solving, individualized goal setting, and personal behavioral change "experiments" designed to help patients set priorities and to become better self-managers of both diabetes and their mood. As part of the intervention activities, group members will be advised to monitor their blood sugar levels, blood pressure, and mood on a daily basis.
  Interventions: Behavioral: Empowerment and CBT Classes

INTERVENTIONS:
Behavioral: Empowerment and CBT Classes — Participants randomized to the intervention arm will receive a manual with 3 CBT modules and 1 Diabetes Empowerment module. CBT Module 1 covers "Understanding Depression and Diabetes", Module 2 "How Thoughts Affect Your Mood and Diabetes Care", Module 3 "How Activities Affect Your Mood and Diabetes Care". The Diabetes Empowerment Module covers topics including the following: food, exercise, medicine, diabetes and your health, social support, communication skills, and community resources.
  Other Names: CBT Classes; Diabetes Classes
  Arms: Empowerment and CBT Classes

SUMMARY:
In this project, investigators examine the impact of a mood treatment enhanced diabetes self-care intervention for depressed, low-income Latino diabetics. The investigators hypothesize that the mood treatment enhancement will lead to significant improvement in both diabetes and depression outcomes as compared with the self-care intervention alone.

DETAILED DESCRIPTION:
The Phase I pilot recruited older Latinos from Dr. Mangione's previous study (who agreed to participate in future research) and 10 participants from a community settings. Those with low mood and poor glycemic control were offered a 12-week intervention combining cognitive behavioral therapy mood management techniques and diabetes self-care into one seamless intervention. Drs. Mangione and Miranda supervised and reviewed (through audiotapes) well-trained health educators conducting the intervention sessions. The study manuals were modified following this Phase I pilot intervention.

The final intervention manual was tested in a randomized trial in Phase II, compared the Mood and Diabetes Empowerment and Improvement Training intervention with enhanced care as usual (providing participants with a letter regarding their mood and hemoglobin (Hb)A1c with recommendations for improving care for their provider). The target population was low-income Latinos with depression and poor glycemic control. Both mood and diabetes outcomes are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Latino men and women age 50 and older
* Must speak English or Spanish
* Hb A1c greater than or equal to 8%
* Currently not taking medication for depression
* A score of 5 or greater on the Geriatric Depression Scale (GDS)

Exclusion Criteria:

* Persons who are legally blind, dialysis dependent, diagnosed with dementia, and/or with hemiparesis from a cerebral vascular accident
* Do not have sufficient hearing or cognitive function

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2009-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Miranda, PhD, Principal Investigator — UCLA Psychr & Biobehav Sci
Locations (1):
- UCLA Psychr & Biobehav Sci, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Empowerment and CBT Classes: Participants will attend weekly 2-hour group Empowerment and CBT classes for 12 weeks led by two trained health educators. Participants will learn cognitive behavioral therapy (CBT) techniques to manage their mood. Then participants will learn a diabetes education format grounded in empowerment theory that employs group problem solving, individualized goal setting, and personal behavioral change "experiments" designed to help patients set priorities and to become better self-managers of both diabetes and their mood. Group members will be advised to monitor their blood sugar levels, blood pressure, and mood on a daily basis.
  Empowerment and CBT Classes: Participants will receive a manual with 3 CBT modules and 1 Diabetes Empowerment module. CBT Module 1 covers "Understanding Depression and Diabetes", Module 2 "How Thoughts Affect Your Mood and Diabetes Care", Module 3 "How Activities Affect Your Mood and Diabetes Care". The Diabetes Empowerment Modu
Period: Overall Study
Arm/Group | Wait-listed Control Group | Empowerment and CBT Classes
Started | 39 | 82
Completed | 27 | 59
Not Completed | 12 | 23
Not completed — Lost to Follow-up | 8 | 18
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wait-listed Control Group | Empowerment and CBT Classes | Total
Number analyzed (Participants) | 39 | 82 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (7.8) | 60 (8.4) | 60 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 57 | 86
  Male | 10 | 25 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  Mexican | 32 | 57 | 89
  Central American | 7 | 25 | 32
Hemoglobin A1c [Mean (Standard Deviation); unit: %] | 10.1 (1.7) | 9.8 (1.7) | 9.9 (1.7)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 79.0 (10.6) | 80.0 (10.8) | 79.4 (10.7)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 137.7 (21.4) | 138.9 (19.4) | 138.5 (20)
Low Density Lipoprotein-C [Mean (Standard Deviation); unit: mg/dL] | 110.3 (32.4) | 109.6 (37.0) | 109.8 (35.5)
Geriatric Depression Scale (GDS) [Mean (Standard Deviation); unit: units on a scale] — The Geriatric Depression Scale (GDS) measures depression in older adults. The short form we used consists of 15 yes or no questions. The scale range is 0 to 15, where higher scores indicate greater severity of depression.
  units on a scale | 6.5 (3.6) | 7.3 (3.9) | 7.1 (3.8)
Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-9 (PHQ-9) measures depression in patients. The questionnaire consists of 9 questions where patients self report how frequently they have depression symptoms over the past two weeks. The scale ranges is 0 to 27 where higher scores indicate greater severity of depression.
  units on a scale | 6.5 (3.6) | 11.1 (5.1) | 10.5 (5.1)
EQ-5D [Mean (Standard Deviation); unit: units on a scale] — The EQ-5D measures general quality of life. The index score is based on 5 questions about mobility, self-care, pain, usual activities, and psychological status. The EuroQol Group provides a U.S. preference-weighted algorithm to calculate the index scores. A score of 1 indicates no problems while a score of -0.11 indicates severe problems.
  The scale score is based on a visual analog of a thermostat, where 0 represents worst imaginable health and 100 represents best imaginable health. Patients mark a tick for where they feel their health is on that scale.
  units on a scale
    Scale Score | 60.2 (19) | 63.6 (13) | 61.3 (17)
    Index Score | 0.655 (0.20) | 0.795 (0.21) | 0.699 (0.21)
Yale Physical Activity Scale - Index Summary Score [Mean (Standard Deviation); unit: units on a scale] — The Yale Physical Activity Scale measures physical function and activities of daily living. Five activity indices (vigorous activity, leisurely walking, moving, standing and sitting) are calculated by multiplying the frequency of activity with the duration and a weighted factor. The 5 indices are then summed to create an index summary. Higher scores indicate more activity. The minimum and maximum scores are 0 and 142.
  units on a scale | 45.8 (28) | 48.3 (28) | 47.5 (28)
Self-Efficacy (Diabetes Empowerment Scale) [Mean (Standard Deviation); unit: units on a scale] — The Diabetes Empowerment Scale Short Form (DES-SF) measures diabetes-related psychosocial self-efficacy. The questionnaire presents 8 statements on self efficacy where participants rate how strongly they agree. The answers are summed to create a score where higher scores indicate more empowerment. The score range is 0 to 8.
  units on a scale | 3.88 (2.6) | 3.72 (2.5) | 3.77 (2.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (5.7) | 32.6 (6.4) | 31.4 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c at 6 Months
Description: Hemoglobin A1c (HbA1c) measures glycemic control over the past three months. HbA1c was measured by a blood draw and laboratory test.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Groups:
- Wait-listed Control Group: Participants in the Wait-listed Control Group received augmented access and communication with a primary care provider. The augmentation consisted of providing the participant with a letter to be shared with their primary care doctor indicating their Hb A1c level and depression score at the time of eligibility screening. The research team also attached a list of local mental health service providers to the letter. The participants randomized to the wait-listed control group will be offered access to the intervention after the trial is completed in the event that the randomized controlled trial (RCT) has significant results.
- Empowerment and CBT Classes: Participants attended weekly 2-hour group Empowerment and CBT classes for 12 weeks led by two trained health educators. Participants learned cognitive behavioral therapy (CBT) techniques to manage their mood. After CBT, participants learned a diabetes education format that is grounded in empowerment theory that employs group problem solving, individualized goal setting, and personal behavioral change "experiments" designed to help patients set priorities and to become better self-managers of both diabetes and their mood. As part of the intervention activities, group members will be advised to monitor their blood sugar levels, blood pressure, and mood on a daily basis.
Arm/Group | Wait-listed Control Group | Empowerment and CBT Classes
Number analyzed (Participants) | 27 | 59
percentage of glycated hemoglobin | -0.7 (1.5) | -1.6 (2.4)

2. Primary Outcome: Change From Baseline in Depression Measures at 6 Months
Description: The Geriatric Depression Scale (GDS) measures depression in older adults. The short form we used consists of 15 yes or no questions. The scale range is 0 to 15, where higher scores indicate greater severity of depression.
  The Patient Health Questionnaire-9 (PHQ-9) measures depression in patients. The questionnaire consists of 9 questions where patients self report how frequently they have depression symptoms over the past two weeks. The scale ranges is 0 to 27 where higher scores indicate greater severity of depression.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wait-listed Control Group | Empowerment and CBT Classes
Number analyzed (Participants) | 28 | 61
units on a scale
  Geriatric Depression Scale | -0.4 (6.6) | -4.7 (4.3)
  Patient Health Questionnaire-9 | 0.4 (4.8) | -6.9 (5.7)

3. Secondary Outcome: Change From Baseline in Blood Pressure at 6 Months
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Wait-listed Control Group | Empowerment and CBT Classes
Number analyzed (Participants) | 27 | 55
mm Hg
  Systolic Blood Pressure | 1.9 (13) | -0.9 (24)
  Diastolic Blood Pressure | 1.30 (7.4) | -1.25 (13)

4. Secondary Outcome: Change From Baseline in Low Density Lipoprotein-C at 6 Months
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Wait-listed Control Group | Empowerment and CBT Classes
Number analyzed (Participants) | 27 | 55
mg/dL | 0.04 (57) | 1.9 (35)

5. Secondary Outcome: Change From Baseline in EQ-5D at 6 Months
Description: The EQ-5D measures general quality of life. The index score is based on 5 questions about mobility, self-care, pain, usual activities, and psychological status. The EuroQol Group provides a U.S. preference-weighted algorithm to calculate the index scores. A score of 1 indicates no problems while a score of -0.11 indicates severe problems.
  The scale score is based on a visual analog of a thermostat, where 0 represents worst imaginable health and 100 represents best imaginable health. Patients mark a tick for where they feel their health is on that scale.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wait-listed Control Group | Empowerment and CBT Classes
Number analyzed (Participants) | 28 | 61
units on a scale
  Scale | 1.75 (19) | 14.7 (21)
  Index Score | -0.02 (0.2) | 0.11 (0.2)

6. Secondary Outcome: Change From Baseline in Yale Physical Activity Scale - Index Summary Score at 6 Months
Description: The Yale Physical Activity Scale measures physical function and activities of daily living. Five activity indices (vigorous activity, leisurely walking, moving, standing and sitting) are calculated by multiplying the frequency of activity with the duration and a weighted factor. The 5 indices are then summed to create an index summary. Higher scores indicate more activity. The minimum and maximum scores are 0 and 142.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wait-listed Control Group | Empowerment and CBT Classes
Number analyzed (Participants) | 28 | 61
units on a scale | -10.5 (28) | 21.5 (34)

7. Secondary Outcome: Change From Baseline in Self-Efficacy (Diabetes Empowerment Scale) at 6 Months
Description: The Diabetes Empowerment Scale Short Form (DES-SF) measures diabetes-related psychosocial self-efficacy. The questionnaire presents 8 statements on self-efficacy where participants rate how strongly they agree. The answers are summed to create a score where higher scores indicate more empowerment. The score range is 0 to 8.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wait-listed Control Group | Empowerment and CBT Classes
Number analyzed (Participants) | 28 | 61
units on a scale | -1.31 (2.9) | 4.31 (2.8)

ADVERSE EVENTS:
Time Frame: Four years
Description: Any suicidality as indicated by self-report, PHQ-9 endorsement of suicidal item, or Geriatric Depression Scale score above 10. Any indication of hyper or hypoglycemia.
Groups:
- Empowerment and CBT Classes: Weekly 2-hour group Empowerment and CBT classes for 12 weeks are led by two trained health educators. Cognitive behavioral therapy (CBT) techniques to manage mood and diabetes education, grounded in empowerment theory that employs group problem solving, individualized goal setting, and personal behavioral change "experiments" designed to help patients set priorities and to become better self-managers of both diabetes and their mood, is presented. Group members monitor their blood sugar levels, blood pressure, and mood on a daily basis. The intervention arm participants receive a manual with 3 CBT modules ("Understanding Depression and Diabetes", "How Thoughts Affect Your Mood and Diabetes Care", and"How Activities Affect Your Mood and Diabetes Care". and 1 Diabetes Empowerment module. covers topics including the following: food, exercise, medicine, diabetes and your health, social support, communication skills, and community resources.
Arm/Group | Wait-listed Control Group | Empowerment and CBT Classes
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/82
Other Adverse Events (participants affected / at risk) | 0/39 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No